CLINICAL TRIAL: NCT02081521
Title: Evaluation of a Multiple Behaviour Programme to Prevent and Manage Diarrhoea Among Children Under-five in Lusaka, Zambia
Brief Title: Evaluation of a Multiple Behaviour Programme for Diarrhoea Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other); Absolute Return for Kids (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: QA511
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Diarrhoeal Disease
Keywords: behaviour change; diarrhoeal disease; handwashing; breastfeeding; diarrhoea management
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community behaviour change campaign (Experimental): Participants will be exposed to the community behaviour change intervention.
  Interventions: Behavioral: Community behaviour change campaign
- No community behaviour change campaign (No Intervention): No community intervention will take place in the control arm, although exposure to some intervention messaging (radio adverts) may take place.

INTERVENTIONS:
Behavioral: Community behaviour change campaign — Community campaign targeting exclusive breastfeeding, handwashing with soap, and use of ORS and zinc to manage child diarrhoea. Includes a range of activities within the community (large events and small group sessions); clinic activities (ORS preparation), radio adverts.
  Arms: Community behaviour change campaign

SUMMARY:
Control of diarrhoeal disease requires a comprehensive package of preventive and curative interventions. in Zambia, the Programme for Awareness and Elimination of Diarrhoea (PAED) aims to reduce child deaths by combating diarrhoea in Lusaka province, Zambia. The behaviour change component of the PAED programme seeks to change behaviours important for diarrhoea prevention (handwashing with soap and exclusive breastfeeding) and improved treatment outcomes (use of oral rehydration solution (ORS) and zinc in home management of child diarrhoea).

The study aims to evaluate the feasibility of implementing a multiple behaviour change community programme to tackle diarrhoeal disease in children under-five and to assess the impact of this programme on practice of the target behaviours by caregivers of children under-five. The research questions will be answered through a a two-arm cluster-randomised trial (eight clusters per study arm).

DETAILED DESCRIPTION:
Specific objectives of the study are as follows:

* Evaluate the effect of the programme on ORS and zinc uptake and usage, exclusive breastfeeding and handwashing with soap (primary objective)
* Determine the extent to which the programme has positively influenced key mediating factors that determine behaviour (i.e. social norms, physical infrastructure, attitudes, and disease and treatment perceptions)
* Investigate which components of the community programme (i.e. specific activities in clinics, community events etc.) are linked to the success of the programme (most acceptable, feasible etc) and in what context

  o Validate model of intervention theory that explains how the context and mechanisms of the intervention interact to produce behavioural outcomes
* Determine which target populations are more likely to uptake the desired behaviours and identify the supporting factors that might explain this
* Conduct process evaluation to assess i) if the programme has been implemented as intended, ii) if the desired levels of reach and coverage have been achieved, iii) costs of implementation, iv) the extent to which changes in behaviour are likely to be due to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* caregiver with child under six months (for assessment of handwashing and exclusive breastfeeding outcomes - healthy volunteers)
* caregiver with child under five years with current or recent (last 7 days) diarrhoea (for assessment of ORS and zinc outcomes)

Exclusion Criteria:

* Not resident in study area

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 640 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in target behaviour: zinc use | six weeks post-intervention
  Proportion of under-five diarrhoeal episodes receiving zinc.
  The study aims to demonstrate the intervention can successfully change behaviour and therefore no health outcomes were chosen and there is a primary outcome for each behaviour.
Change in target behaviour: correct ORS preparation | six weeks post-intervention
  Proportion of caregivers able to demonstrate correct ORS preparation.
Change in target behaviour: Exclusive breastfeeding | six weeks post-intervention
  Proportion of mothers exclusively breastfeeding infants 0-5 months of age.
Change in target behaviour: Handwashing with soap | six weeks post-intervention
  Proportion of observed handwashing events where there is risk of faecal contamination (i.e. after latrine and when dealing with child stools) accompanied by handwashing with soap

SECONDARY OUTCOMES:
Change in target behaviours: ORS use | six weeks post-intervention
  Proportion of under-five diarrhoeal episodes receiving ORS.
Change in target behaviours: ORS storage | six weeks post-intervention
  Proportion of caregivers storing ORS sachets at home
Change in target behaviours: zinc trial | six weeks post-intervention
  Proportion of caregivers of a child under-five who have ever used zinc to treat diarrhoea in a child
Zinc awareness | six weeks post-intervention
  Proportion of caregivers who have heard of zinc for diarrhoea treatment
Change in target behaviours: exclusive breastfeeding 0-2 months | six weeks post-intervention
  Proportion of mothers exclusively breastfeeding infants 0-2 months of age.
Change in target behaviours: predominant breastfeeding | six weeks post-intervention
  Proportion of mothers predominantly breastfeeding infants 0-5 months of age.
Change in target behaviours: handwashing with soap at key times | six weeks post-intervention
  Proportion of observed handwashing events associated with food handling or faeces accompanied by handwashing with soap
Change in target behaviours: use of soap | six weeks post-intervention
  Proportion of observed handwashing occasions where soap is used

CONTACTS AND LOCATIONS:
Overall Officials: Roma Chilengi, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (1):
- Centre for Infectious Disease Research Zambia, Lusaka, Lusaka Province, Zambia

REFERENCES:
- [Derived] Greenland K, Chipungu J, Chilekwa J, Chilengi R, Curtis V. Disentangling the effects of a multiple behaviour change intervention for diarrhoea control in Zambia: a theory-based process evaluation. Global Health. 2017 Oct 17;13(1):78. doi: 10.1186/s12992-017-0302-0. PMID 29041941
- [Derived] Greenland K, Chipungu J, Curtis V, Schmidt WP, Siwale Z, Mudenda M, Chilekwa J, Lewis JJ, Chilengi R. Multiple behaviour change intervention for diarrhoea control in Lusaka, Zambia: a cluster randomised trial. Lancet Glob Health. 2016 Dec;4(12):e966-e977. doi: 10.1016/S2214-109X(16)30262-5. PMID 27855872